CLINICAL TRIAL: NCT03254004
Title: Postoperative Pembrolizumab for the Patients Who Have Solid Predominant or Micropapillary Lung Adenocarcinoma With Pathologic Stage I and Primary Tumor Than 4 cm
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jhingook Kim, MD, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-08-032
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Lung Adenocarcinoma, Stage I
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Pembrolizumab 200mg injection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm: pembrolizumab (Experimental): pembrolizumab 200 mg every 3 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — pembrolizumab 200 mg every 3 weeks till 1 year or disease recurrence or intolerable toxicity.

SUMMARY:
A single center, open-label, single arm study in patients who have solid or micropapillary adenocarcinoma with pathologic stage I and primary tumor no more than 4 cm. Pembrolizumab 200 mg every 3 weeks

DETAILED DESCRIPTION:
This is a single center, open-label, single arm study in patients who have solid or micropapillary adenocarcinoma with pathologic stage I and primary tumor no more than 4 cm. Patients will be treated with pembrolizumab 200 mg every 3 weeks till 1 year or disease recurrence or intolerable toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Primary lung adenocarcinoma patients with stage I and less than 4 centimeter of primary tumor, whose tumor should be solid-predominant or micropapillary (>5%) by postsurgical pathological examination.

   * Note: The specific methods and principles of pathology results follow the WHO's pathology guidelines. The institution uses diagnostic pathology results from the institution.
   * Note: Adenocarcinoma, solid-predominant subtype; This variant shows a major component of polygonal tumor cells forming sheets that lack recognizable patterns of adenocarcinoma, i.e., acinar, papillary, micropapillary, or lepidic growth. If the tumor is 100% solid, intracellular mucin should be present in >5 tumor cells in each of two high-power fields, and confirmed with histochemical stains for mucin.
   * Note: Adenocarcinoma, micropapillary subtype; This variant has, as a major component, tumor cells growing in papillary tufts forming florets that lack fibrovascular cores. These may appear detached from and/or connected to alveolar walls. The tumor cells are usually small and cuboidal, with variable nuclear atypia. Ring-like glandular structures may float within alveolar spaces. Vascular and stromal invasion is common. Psammoma bodies may be seen.
2. Be willing and able to provide written informed consent/assent for the trial.
3. No evidence of disease (NED) after surgical resection on baseline tumor imaging (chest CT, covering up to both adrenals). The following conditions are satisfied with the condition of the complete ablation(R0):

   * free resection margins proved microscopically
   * no evidence of nodal metastasis by ststematic and radical nodal dissection
4. Be 20 years of age on day of signing informed consent.
5. Be willing to provide tissue from surgical specimen or excisional biopsy of a tumor lesion.
6. Have a performance status of 0 or 1 on the ECOG Performance Scale.
7. Demonstrate adequate organ function as defined in Table 1, all screening labs should be performed within 10 days of treatment initiation.

   Table 1 Adequate Organ Function Laboratory Values
   * Hematological

     * Absolute neutrophil count (ANC): ≥1,500 /mcL
     * Platelets: ≥100,000 / mcL
     * Hemoglobin: ≥9 g/dL or ≥5.6 mmol/L without transfusion or EPO dependency (within 7 days of assessment)
   * Renal

     * Serum creatinine OR Measured or calculateda creatinine: ≤ 1.5 X upper limit of normal (ULN) OR
     * clearance(GFR can also be used in place of creatinine or CrCl): ≥ 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
   * Hepatic

     * Serum total bilirubin: ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
     * AST (SGOT) and ALT (SGPT): ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases
     * Albumin: >2.5 mg/dL
   * Coagulation

     * International Normalized Ratio (INR) or Prothrombin Time (PT): ≤ 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intenede use of anticoagulants
     * Activated Partial Thromboplastin Time (aPTT): ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intenede use of anticoagulants
     * Creatinine clearance should be calculated per institutional standard.
8. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

   * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
10. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

    * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Is on chronic systemic steroids. Subjects with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study.
3. Hypersensitivity to pembrolizumab or any of its excipients.
4. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
7. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
8. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
9. Has known history of, or any evidence of active, non-infectious pneumonitis.
10. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
17. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy.

    * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-10-08 (Actual); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
To assess the improvement of disease-free survival rate by adjuvant therapy with pembrolizumab for solid or micropapillary adenocarcinoma with pathologic stage I and tumor size no more than 4 cm. | up to 16 times. (screening, every 4 cycles during the study, every 3 months till 1 year since the study treatment, and then every 4 months afterward till 2 years and thereafter every 6 months till 3 years)
  RECIST V1.1

CONTACTS AND LOCATIONS:
Overall Officials: jhingook Kim, MD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical centre, Seoul, Kangnam, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim J, Bang YH, Park S, Jung HA, Sun JM, Ahn JS, Ahn MJ, Jeon YJ, Lee J, Cho JH, Kim HK, Choi YS, Zo JI, Shim YM, Kang JH, Lee J, Choi YL, Han J, Hwang S, Lee HY, Lee SH. Adjuvant pembrolizumab therapy for completely resected stage I lung adenocarcinoma with micropapillary or solid histological subtypes: a single-center, single-arm, phase 2 trial. EClinicalMedicine. 2025 Jun 4;84:103282. doi: 10.1016/j.eclinm.2025.103282. eCollection 2025 Jun. PMID 40524802